CLINICAL TRIAL: NCT03618784
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-controlled Phase I/2a Clinical Trial to Evaluate the Efficacy and Safety of FURESTEM-RA Inj. for Moderate to Severe Rheumatoid Arthritis
Brief Title: Safety and Efficacy of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K0202
Record Dates: First submitted 2018-07-24; First posted 2018-08-07 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis
Keywords: FURESTEM-RA Inj.; Rheumatoid Arthritis; Cell therapy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FURESTEM-RA Inj. (Experimental)
  Interventions: Biological: FURESTEM-RA Inj
- Placebo Comparator: Placebo (Placebo Comparator)
  Interventions: Other: sterile saline

INTERVENTIONS:
Biological: FURESTEM-RA Inj — The allogeneic umbilical cord blood-derived mesenchymal stem cells of each dose level as below were mixed into an IV bag containing 100 ml of sterile saline solution and the IV bag was gently massaged to obtain homogeneous mixture of the cell suspension.
  Administer the constituted cell suspension by IV infusion to a subject. The infusion should be completed in 60 minutes using infusion pump.
  * Dose level 1: 5.0 x 10^7 cells /body 3 repeated intravenous injection at 4 week intervals
  * Dose level 2: 1.0 x 10^8 cells /body 3 repeated intravenous injection at 4 week intervals
  Arms: FURESTEM-RA Inj.
Other: sterile saline — sterile saline 3 repeated intravenous injection at 4 week intervals
  Placebo were mixed into an IV bag containing 100 ml of sterile saline solution and the IV bag was gently massaged to obtain homogeneous mixture of the cell suspension.
  Administer the constituted cell suspension by IV infusion to a subject. The infusion should be completed in 60 minutes using infusion pump.
  Arms: Placebo Comparator: Placebo

SUMMARY:
Safety and Efficacy of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid arthritis

DETAILED DESCRIPTION:
Phase 1: Single center, open Phase 2a : Multi-center, randomized, double-blind, parallel, placebo Clinical Trial to Evaluate the Efficacy and Safety of FURESTEM-RA Inj. for Moderate to Severe Rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

1. of either gender, 19-80years old
2. Subjects must be diagnosed according to the 2010 ACR/EULAR criteria for at least 12 weeks duration.
3. Subjects must be diagnosed with ACR functional class I. II, III
4. ≥ 6 tender joints, swollen joints (68 joint count) at Screening
5. Subject who has moderate to severe disease activity (DAS28-ESR>3.2) on screening visit
6. History of treatment for one of conventional DMARDs or biologic DMARDs or JAK inhibitors AND people diagnosed with either (a) or (b) by a trained person, or people that have potential side effects thus not qualified from using biologic DMARDs.

   1. people that have no effect with permitted dose taking for more than 3 months
   2. people with a history of side effects of relevant treatment
7. Subjects must be taking cDMARDs(including methotrexate, sulfasalazine, hydroxychloroquine, leflunomide) or tacrolimus of stable dose More than 12 weeks before baseline visit and be willing to remain on stable dose throughout the study
8. If subject is currently administering steroids everyday, when steroid dose is converted into prednisolone oral dose, the subject should take a stable dose(≤10mg/day) over 4 weeks on screening visit
9. In case of taking NASAIDs, Tramadol patients with stable amount of medication at least 2 weeks before screening visit.
10. During screening visit , patients with an ESR result of 28mm/hr; patients with a 1.0mg/dL or greater in a CRP testing
11. Subject who understands and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects who is diagnosed ACR function class IV Rheumatoid Arthritis
2. Patients who are judged by the PI(or Sub-I) to be unable to participate in clinical trials due to uncontrolled or unstable cardiovascular disease or severe blood disease
3. Subjects who has AIDS, other rheumatic disease(Crohn's disease, systemic lupus erythematosus, lyme disease, psoriatic arthritis, spondylarthropathy, infectious or reactive arthritis, reiter's syndrome, etc.)
4. Prior use of bDMARDs, within the following windows prior to baseline

   * 24 weeks for Rituximab
   * 10 weeks for Abatacept, Golimumab, Certolizumab pegol, Tocilizumab
   * 7 weeks for Infliximab
   * 4 weeks for Etanercept
   * 3 weeks for Tofacitinib, Baricitinib
5. Subject who has history of hypersensitivity, heavy metal poisoning, etc. to drugs which is composed of similar components.
6. Subject who has treated intravenous, intramuscular steroid injection within 2 weeks before screening visit or intra-articular steroid injection within 4 weeks before screening visit
7. Subject who has administered ACTH(adrenocorticotropic hormone) agents within 4 weeks before screening visit
8. Subject who has undergone administration of any investigational drug within 30 days before screening visit.
9. Use of prohibited medication or inability to avoid the use of prohibited medication during the study
10. Pregnant, breast-feeding women
11. A female or male in their childbearing ages that is not willing to take proper contraceptive methods during a study
12. Subject who has sever dyshepatia (Serum creatinine level ≥ 1.7mg/dl)
13. Subject who has severe renal dysfunction (ALT/AST/bilirubin value ≥ 2 upper limit of the normal range at screening test)
14. Any other condition which the PI Judges would make patient unsuitable for study participation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Safety of FURESTEM-RA Inj. - number of adverse events | 4 weeks follow-up after treatment
  Evaluate the number of adverse events Safety of FURESTEM-RA Inj.

SECONDARY OUTCOMES:
Efficacy as measured by ACR(American College of Rheumatology)20,50,70 reaction rate | 16 weeks follow-up after treatment
Efficacy as measured by EULAR (European League Against Rheumatism)reaction rate | 16 weeks follow-up after treatment
Efficacy as measured by DAS(Disease activity scores)28-ESR | 16 weeks follow-up after treatment
  DAS range is from ≥ 3.2 (inactive) , >3.2 but ≤ 5.1(moderate), >5.1(very active)
Efficacy as measured by KHAQ(Korean Health assessment questionnaire) | 16 weeks follow-up after treatment
  KHAQ range is from 0 (clear) to 60 (severe)
Efficacy as measured by CDAI (clinical disease activity index) | 16 weeks follow-up after treatment
  CDAI range is from 0 (clear) to 76 (severe)
Efficacy as measured by 100mm Pain VAS(Visual analogue scale) | 16 weeks follow-up after treatment
  100mm Pain VAS range is from 0 (clear) to 100 (severe)
Total number of use and consumed amount of rescue medicine | 16 weeks follow-up after treatment
Change in Cytokine(TNF-a, Interleukin (IL)-1b, IL-4,IL-6,IL-8,IL-10,IL-13,IL-17A,IL-21,IL-22) | 16 weeks follow-up after treatment

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Chonnam National University Hospital, Gwangju
  - Gangdong Kyung Hee University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul Hospital attached to Soonchunhyang University, Seoul
  - Seoul national University Boramae, Seoul
  - Seoul National University Hospital, Seoul